CLINICAL TRIAL: NCT03186703
Title: Evaluating the Impact of the McMaster Optimal Aging Portal on Knowledge, Behavioural Intentions and Health Behaviours Related to Cancer Risk in Underserved Populations.
Brief Title: Evaluating the Impact of the McMaster Optimal Aging Portal on Cancer Prevention Behaviours in Underserved Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 316590
Record Dates: First submitted 2017-04-07; First posted 2017-06-14 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2019-03

CONDITIONS: Cancer
Keywords: Cancer prevention; Knowledge translation; Physical activity; Diet; Alcohol; Smoking
MeSH Terms: conditions — Neoplasms; Motor Activity; Smoking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored knowledge translation (Experimental): During the 12-week intervention, intervention group participants will have access to the Portal and will receive targeted weekly email alerts including blog posts and evidence summaries relevant to cancer prevention and be invited to follow a Twitter and Facebook feed; a unique hashtag will be created to identify and collate relevant cancer prevention information.
  Interventions: Behavioral: Tailored knowledge translation
- Control (No Intervention): Participants in the control group will have access to the Portal in a 'self-serve' fashion. These participants will be able to browse the Portal, subscribe to email alerts, follow social media, etc. but will not receive the tailored intervention.

INTERVENTIONS:
Behavioral: Tailored knowledge translation — Tailored knowledge translation strategies specific to evidence-based cancer prevention recommendations
  Arms: Tailored knowledge translation

SUMMARY:
The goal of the McMaster Optimal Aging Portal is to be a trustworthy source for health information. The Portal team can see (through measuring analytics of website use) that thousands of people are using the Portal and the knowledge-sharing strategies in place (email alerts, Twitter and Facebook), with many more users added each month. Previous studies have measured the quality and trustworthiness of health information available online; others have studied the numbers and populations who use different types of information and how easy it is to use and understand. This study builds on that knowledge to find out: if easy-to-understand evidence-based messages reach members of the public, do these messages change what people know and think to do to stay healthy (in this case, what they know and think to do to lower their risk of cancer)?

DETAILED DESCRIPTION:
Half of cancers are preventable through lifestyle modification such as smoking cessation, healthy eating, increasing physical activity and reducing alcohol intake; however, few Canadians engage in behaviours that are in line with cancer prevention guidelines. This may be in part due to lack of access to evidence-based information and the mixed messages on effective cancer prevention strategies that are propagated in the popular media.

The McMaster Optimal Aging Portal (the Portal) is a knowledge translation (KT) tool launched in 2014 to increase public access to trustworthy health information. Citizen-friendly content (blog posts, evidence summaries, web resource ratings) provide easy-to-read 'bottom line' messages appropriate for all audiences. Investigators would now like to know if and how KT strategies used to disseminate citizen-targeted information on cancer prevention impact knowledge, behavioural intentions and health behaviours of Canadian adults.

This study will use a sequential mixed-methods design consisting of a two-arm randomized controlled trial (RCT) and a qualitative process study to explore RCT findings in depth. This formative approach will allow for a deeper analysis of the outcomes of interest (knowledge, intentions and behaviours), and the KT process. Following baseline data collection, eligible participants will be randomized to a 12-week intervention or control group.

During the intervention, participants will have access to the Portal, be invited to follow a Twitter and Facebook feed, and receive tailored weekly email alerts including blog posts and evidence summaries on cancer prevention. Control group participants will have access the Portal in a 'self-serve' fashion, but will not receive KT strategies.

ELIGIBILITY:
Inclusion Criteria:

* English speaking

Exclusion Criteria:

* Previous cancer diagnosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Website engagement | 12 weeks
  Number of clicks
Email engagement | 12 weeks
  Number of clicks
Social media engagement | 12 weeks
  Number of clicks

SECONDARY OUTCOMES:
Knowledge questionnaire | 12 weeks, 3-months post-intervention
  Participants knowledge of cancer prevention recommendations and guidelines
Beliefs questionnaire | 12 weeks, 3-months post-intervention
  Participants beliefs about the importance of lifestyle in prevention cancer
Intentions questionnaire | 12 weeks, 3-months post-intervention
  Participants intentions to engage in lifestyle behaviours in line with cancer prevention guidelines
Godin leisure time exercise questionnaire | 12 weeks, 3 months post-intervention
  Physical activity
Dietary Screener Questionnaire | 12 weeks, 3 months post-intervention
  Dietary intake
Tobacco Questions for Surveys, World Health Organization | 12 weeks, 3 months post-intervention
  Current smoking behaviour
Seven-day recall alcohol | 12 weeks, 3 months post-intervention
  Alcohol intake
Participant satisfaction | 12 weeks
  Collected using qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Dobbins, RN, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neil-Sztramko SE, Belita E, Levinson AJ, Boyko J, Dobbins M. Evaluation of an online knowledge translation intervention to promote cancer risk reduction behaviours: findings from a randomized controlled trial. BMC Cancer. 2019 Nov 21;19(1):1138. doi: 10.1186/s12885-019-6361-2. PMID 31752751